CLINICAL TRIAL: NCT00655343
Title: GvHD Prophylaxis With ATG-Fresenius S in Allogeneic Stem Cell Transplantation From Matched Unrelated Donors: A Randomized Phase III Multicenter Trial Comparing a Standard GvHD Prophylaxis With Cyclosporine A and Methotrexate With Additional Pretransplant ATG-Fresenius S
Brief Title: Acute Graft-Versus-Host Disease (aGvHD) Prophylaxis With ATG-Fresenius in Matched Unrelated Donor-Stem Cell Transplantation (MUD-SCT)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Neovii Biotech (Industry)
Collaborators: University Medical Center Freiburg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AP-AS-21-DE
Record Dates: First submitted 2008-04-03; First posted 2008-04-09 (Estimated); Last update posted 2011-12-12 (Estimated); Status verified 2011-12

CONDITIONS: Graft vs Host Disease
Keywords: GvHD; aGvHD prophylaxis; Matched unrelated donor; ATG; SCT; BMT; polyclonal antibody; GvHD prophylaxis for patients with ALL, AML, CML, MDS, OMF; Patients with allogeneic BM or PBSC transplantation; Patients with a matched unrelated donor
MeSH Terms: conditions — Graft vs Host Disease; Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ATG-F (Experimental): ATG-Fresenius S (20 mg/kg body weight at days -3 to -1 (total dose: 60 mg/kg)
  cyclosporine A (target trough level > 200ng/ml (day -1 until day +100)
  methotrexate: 15mg/m2 at day +1, 10mg/m2 at days +3, +6, and +11
  Interventions: Drug: ATG-Fresenius S
- non-ATG-F (No Intervention): cyclosporine A (target trough level > 200ng/ml (day -1 until day +100)
  methotrexate: 15mg/m2 at day +1, 10mg/m2 at days +3, +6, and +11

INTERVENTIONS:
Drug: ATG-Fresenius S — 20 mg rabbit immunoglobulin (IgG) in 1 ml of sterile solution
  20 mg/kg body weight per day diluted in 500 ml physiological saline, slow intravenous infusion at days -3, -2, -1 prior to transplantation
  Other Names: ATG-Fresenius; Anti-T-Lymphocyte globulin
  Arms: ATG-F

SUMMARY:
The study aim is to evaluate the influence of the anti-T-lymphocyte globulin ATG-Fresenius S given pre-transplant in addition to standard GvHD prophylaxis with cyclosporine A and a short course of methotrexate with respect to efficacy and safety.

DETAILED DESCRIPTION:
To assess the efficacy of ATG-FRESENIUS S in addition to standard therapy (cyclosporine A / methotrexate) with respect to early treatment failure defined by the occurrence of severe acute GvHD grade III-IV or early mortality within 100 days post transplantation compared to standard therapy alone.

All patients receive myeloablative therapy. Recommended regimens: For patients with ALL: fractionated TBI (8-12 Gy) plus cyclophosphamide (1-2 x 60 mg/kg) [etoposide/melfalan are also allowed]. For all other indications: either TBI (8-12 Gy) or busulfan (per os 14-16 mg/kg b.w. or equivalent for IV administration) plus cyclophosphamide (1-2 x 60 mg/kg) or thiotepa ≥ 15 mg/kg or BCNU ≥ 300 mg/m2.

Conditioning regimens may differ from centre to centre; each centre decides for constant (disease specific) regimen(s) throughout the whole study period.

Standard GvHD prophylaxis consists of cyclosporine A (target trough level ≥ 200 ng/ml starting from day -1 until day +100) and short course methotrexate (15 mg/m2 at day +1, 10 mg/m2 at days +3, +6 and +11).

ELIGIBILITY:
Inclusion Criteria:

Participation of patients in simultaneous diagnostic and comprehensive therapeutical trials for certain entities is allowed.

* Patients 18-60 years of age;
* Patients suffering from one of the following diseases:

  * AML: 1st complete remission (CR1) or beyond 1st remission (CR2, CR3), in relapse, not in remission (primary refractory, induction failure);
  * ALL: 1st complete remission (CR1) or beyond 1st remission (CR2, CR3), in relapse, not in remission (primary refractory, induction failure);
  * MDS, if transplantation is medically indicated: RA (with poor risk factors as classified by the International Prognostic Scoring System of MDS), RARS, RAEB, RAEB-t, CMML;
  * CML: beyond 1st chronic phase (CP1): accelerated phase, blast crisis, chronic phase (CP2, CP3);
  * OMF, if transplantation is medically indicated: Osteomyelofibrosis;
* Patients designated to undergo allogeneic bone marrow transplantation or allogeneic peripheral blood stem cell transplantation;
* Patients with a HLA-A, -B (DNA-based, 2 digits), HLA-DRB1, -DQB1 (DNA-based 4 digits) matched (8 out of 8 alleles) unrelated donor; serological typing is not required
* Patients with a Karnofsky Performance Score (KPS): > 60%;
* Patients who underwent all obligatory screening examinations (special examinations within the last 4 weeks);
* Patients who have given their written informed consent to participate in the study.

Exclusion Criteria:

* Patients with significant cardiac (e.g. ejection fraction <50%), pulmonary (e.g. FEV1 <50%), renal (e.g. creatinine > 1.5 mg/dl), metabolic (e.g. bilirubin > 2.0 mg/dl) and/or CNS disease, currently uncontrolled by treatment, which may interfere with the completion of the study;
* Patients with any bacterial, viral, or fungal infections not under adequate antimicrobial control;
* Patients who are known to have serum hepatitis or who are carriers of the Hepatitis B surface antigen (HBs-Ag), or Hepatitis C antibody, or who are known to have a positive result to the test of HIV antibodies;
* Patients with any additional concurrent or previous malignant disease;
* Patients with known hypersensitivity to rabbit immunoglobulin antibodies in past patient history or with known allergy to any substance chemically related to the study medication;
* Pregnant (β-HCG test) or lactating women;
* Patients who formerly underwent transplantation including previous autologous transplants;
* Patients who cannot communicate reliably with the investigator or who are not likely to cope with the requirements of the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 202 (Actual)
Dates: Start 2003-02; Primary Completion 2007-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Primary: Early treatment failure defined by the occurrence of severe acute GvHD (°III-°IV) or early mortality within 100 days post transplantation. | 100 days

SECONDARY OUTCOMES:
Time to onset of acute GvHD, incidence and severity of infections until day +100, time to engraftment, incidence of cGvHD, disease free survival, relapse, death without relapse, overall survival, safety, tolerability. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Juergen Finke, Prof. Dr., Principal Investigator — Albert-Ludwigs-University Freiburg
Locations (1):
- Universität Freiburg, Medizinische Klinik, Abteilung Innere Medizin I, Hämatologie/Onkologie, Freiburg im Breisgau, Baden-Wurttemberg, Germany

REFERENCES:
- [Result] Socie G, Schmoor C, Bethge WA, Ottinger HD, Stelljes M, Zander AR, Volin L, Ruutu T, Heim DA, Schwerdtfeger R, Kolbe K, Mayer J, Maertens JA, Linkesch W, Holler E, Koza V, Bornhauser M, Einsele H, Kolb HJ, Bertz H, Egger M, Grishina O, Finke J; ATG-Fresenius Trial Group. Chronic graft-versus-host disease: long-term results from a randomized trial on graft-versus-host disease prophylaxis with or without anti-T-cell globulin ATG-Fresenius. Blood. 2011 Jun 9;117(23):6375-82. doi: 10.1182/blood-2011-01-329821. Epub 2011 Apr 5. PMID 21467544
- [Result] Finke J, Bethge WA, Schmoor C, Ottinger HD, Stelljes M, Zander AR, Volin L, Ruutu T, Heim DA, Schwerdtfeger R, Kolbe K, Mayer J, Maertens JA, Linkesch W, Holler E, Koza V, Bornhauser M, Einsele H, Kolb HJ, Bertz H, Egger M, Grishina O, Socie G; ATG-Fresenius Trial Group. Standard graft-versus-host disease prophylaxis with or without anti-T-cell globulin in haematopoietic cell transplantation from matched unrelated donors: a randomised, open-label, multicentre phase 3 trial. Lancet Oncol. 2009 Sep;10(9):855-64. doi: 10.1016/S1470-2045(09)70225-6. Epub 2009 Aug 18. PMID 19695955
- [Derived] Chakupurakal G, Freudenberger P, Skoetz N, Ahr H, Theurich S. Polyclonal anti-thymocyte globulins for the prophylaxis of graft-versus-host disease after allogeneic stem cell or bone marrow transplantation in adults. Cochrane Database Syst Rev. 2023 Jun 21;6(6):CD009159. doi: 10.1002/14651858.CD009159.pub3. PMID 37341189
- [Derived] Finke J, Schmoor C, Bethge WA, Ottinger H, Stelljes M, Volin L, Heim D, Bertz H, Grishina O, Socie G. Long-term outcomes after standard graft-versus-host disease prophylaxis with or without anti-human-T-lymphocyte immunoglobulin in haemopoietic cell transplantation from matched unrelated donors: final results of a randomised controlled trial. Lancet Haematol. 2017 Jun;4(6):e293-e301. doi: 10.1016/S2352-3026(17)30081-9. PMID 28583289